CLINICAL TRIAL: NCT06797362
Title: Expanded Access Treatment of Zidesamtinib (NVL-520) in Patients With Advanced ROS1+ NSCLC or Other ROS1+ Solid Tumors
Brief Title: Expanded Access Program of Zidesamtinib (NVL-520) for Patients With Advanced ROS1+ NSCLC or Other ROS1+ Solid Tumors
Status: Available | Type: Expanded Access
Sponsor: Nuvalent Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NVL-520-EAP
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer; ROS1-positive Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: NVL-520 — Oral tablet
  Other Names: Zidesamtinib

SUMMARY:
The Expanded Access Program will provide an alternate mechanism for these patients, who lack satisfactory therapeutic alternatives and cannot participate in a zidesamtinib clinical trial, to access investigational zidesamtinib.

DETAILED DESCRIPTION:
The purpose of this Expanded Access Program is to provide access to zidesamtinib (NVL-520) an investigational therapy for eligible patients with ROS1 fusion-positive advanced non- small cell lung cancer (ROS1+ NSCLC) who have previously received ≥ 1 prior ROS1 tyrosine kinase inhibitor (TKI) or eligible patients with other ROS1-positive solid tumors who have previously received any prior commercially-available or investigational therapy, and lack satisfactory therapeutic alternatives and are unable to access zidesamtinib through a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Histologically or cytologically confirmed locally advanced or metastatic NSCLC or other solid tumor with documented ROS1 rearrangement.
3. Previously received at least 1 prior ROS1 TKI, with no comparable or satisfactory alternative treatment options, in the opinion of the treating physician.
4. Enrollment in a clinical trial of zidesamtinib is not possible.
5. Adequate organ function and bone marrow reserve.

Exclusion Criteria:

1. Prior receipt of zidesamtinib.
2. Previous surgery, chemotherapy, radiotherapy or other anti-cancer therapy or participation in other studies within timeframe indicated in the protocol.
3. Ongoing anti-cancer therapy.
4. Eligible for ongoing clinical trial with zidesamtinib

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (34):
- United States (6):
  - University of Colorado Anschutz School of Medicine, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, Manhattan, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Washington / Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (2):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Hospital, Toronto, Ontario
- France (4):
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - GCS IUCT Oncopole, Toulouse, Occitanie
  - CHU de Nantes, Nantes, Pays de la Loire Region
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- Italy (6):
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - L'Istituto Europeo di Oncologia S.r.l., Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IRCCS Istituto Oncologico Veneto, Padua
  - AUSL della Romagna - Ravenna, Ravenna
  - Istituto Nazionale Tumori "Regina Elena, Roma
- Netherlands (3):
  - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Netherlands Cancer Institute: NKI, Amsterdam
  - University Medical Center Groningen, Groningen
- Singapore (2):
  - National University Hospital Singapore, Singapore
  - National Cancer Centre Singapore, Singapore
- Spain (4):
  - Uomi Cancer Center-Clinica Tres Torres, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Gregorio Marañón General University Hospital, Madrid
  - Hospital Univ Doce de Octubre, Madrid
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (3):
  - The Royal Marsden Hospital, Sutton, Surrey
  - The Royal Marsden Hospital, London
  - The Christie Hospital, Manchester